CLINICAL TRIAL: NCT00904020
Title: A Prospective, Open-Label, Multicenter Study of the Effectiveness And Safety Of Lidoderm® As Add-On Treatment in Patients With Postherpetic Neuralgia, Diabetic Neuropathy, or Low Back Pain
Brief Title: A Study of the Effectiveness And Safety Of Lidoderm® As Add-On Treatment in Patients With Postherpetic Neuralgia, Diabetic Neuropathy, or Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3220-008
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Postherpetic Neuralgia; Diabetic Neuropathy; Low Back Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Diabetic Neuropathies; Low Back Pain | interventions — Lidoderm

ARMS (1):
- (1) Lidoderm (Experimental): (1) Commercially available Lidoderm (lidocaine patch 5%) was provided to patients with up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain.
  Interventions: Drug: Lidoderm

INTERVENTIONS:
Drug: Lidoderm — Patients participated in a 2-week treatment period. Commercially available Lidoderm (lidocaine patch 5%) was provided to patients with up to four patches applied topically once daily (q24h) to the area of maximal peripheral pain.
  Other Names: Lidocaine patach 5%

SUMMARY:
Patients with a diagnosis of postherpetic neuralgia (PHN), diabetic neuropathy (DN), or low back pain (LBP) who were currently receiving an analgesic regimen that contained gabapentin participated in a Phase IV clinical trial to assess the effectiveness of Lidoderm® administered once daily (q24h) after 14 day in the treatment of PHN, DN, or LBP in patients who had a partial response to a regimen containing gabapentin.

ELIGIBILITY:
Inclusion Criteria:

* Were currently receiving an analgesic regimen that contained gabapentin
* Had been on a stable dose of gabapentin for at least 14 days (same dose ±10% for 14 days)
* Had a partial response to a gabapentin-containing analgesic regimen defined as an average daily pain intensity score of >4 on a ) to 10 scale, with 0 being no pain and 10 being pain as bas as the patients have ever imagined (Question 5 of the Brief Pain Inventory [BPI] within 24 hours prior to the screening visit
* For diabetic patients, had a hemoglobin A1c level <0.13 (normal range, 0.047-0.064)

Exclusion Criteria:

* Had a neurological condition other than that associated with their pain diagnosis that, in the opinion of the investigator, would have interfered with their ability to participate in the study
* Had received an epidural steroid/local anesthetic injection within 14 days prior to study entry
* Had received trigger point injections within 14 days prior to study entry
* Had received Botox injections within 3 months prior to study entry
* Were taking a lidocaine-containing product that could not be discontinued while receiving Lidoderm
* Were taking Class 1 anti-arrhythmic drugs (e.g., mexiletine, tocainide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2002-06; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Average daily pain intensity (Brief Pain Inventory [BPI] Questions 3, 4, 5, and 6) | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)

SECONDARY OUTCOMES:
Pain quality using the Neuropathic Pain Scale (NPS) | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
Investigator and Patient Global Impression of Change | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
Extent of numbness at the site of pain using the Numbness Questionnaire | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
Patient Global Assessment of Pain Relief | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
Safety assessments included Adverse Events (AE), discontinuation due to AEs, physical and neurological examination results, vital signs, clinical laboratory data, sensory testing, numbness testing, and dermal assessments | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
QoL: Pain interference (BPI Question 9) | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)
QoL: Patient Global Assessment of Patch Satisfaction | Visits - V2 (Day 0), V3 (Day 7), V4/EOS (Day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (11):
- United States (11):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Plantation, Florida
  - Marietta, Georgia
  - Burr Ridge, Illinois
  - Overland Park, Kansas
  - Hackensack, New Jersey
  - Altoona, Pennsylvania
  - Cudahy, Wisconsin
  - Greenfield, Wisconsin
  - West Bend, Wisconsin